CLINICAL TRIAL: NCT07280741
Title: Efficacy, Immunogenicity, and Safety of the Recombinant Herpes Zoster Vaccine (RZV) in Patients With Autoimmune Rheumatic Diseases Under Immunomodulators
Brief Title: Recombinant Herpes Zoster Vaccine in Patients With Autoimmune Rheumatic Diseases Under Immunomodulators
Acronym: IMUNO-RZV
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 94187625300000068
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Rheumatic Diseases
Keywords: Immunogenicity; Hepers Zoster; Vaccine; Safety; Immunomodulators; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunomodulator Monotherapy (Experimental): Participants with autoimmune rheumatic diseases who are clinically stable and receiving monotherapy with hydroxychloroquine or sulfasalazine will receive two doses of the recombinant zoster vaccine (RZV, Shingrix) administered intramuscularly on Day 0 and Day 42. Immunogenicity will be evaluated through anti-glycoprotein E antibody titers at baseline, six weeks, and one year after vaccination. Safety, disease activity, and incidence of herpes zoster will be monitored throughout follow-up.
  Interventions: Biological: Recombinant Zoster Vaccine (RZV)

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine (RZV) — VRZ (Shingrix®) is composed of 50 μg of recombinant VZV glycoprotein E (gE) and the liposome-based AS01B (HZ/su) adjuvant system (containing 50 μg of 3-O-desacyl-4'-monophosphoryl lipid A [MPL] and 50 μg of Quillaja saponaria Molina, fraction 21 (QS21), licensed by GSK from Antigenics, a subsidiary of Agenus). Two doses of the vaccine will be administered (0.5 mL) into the deltoid muscle on days (D) 0 and D42.

SUMMARY:
This interventional phase IV clinical trial will evaluate the efficacy, immunogenicity and safety of the adjuvanted recombinant herpes zoster vaccine (RZV) in adults with autoimmune rheumatic diseases (ARDs) receiving immunomodulatory monotherapy. Humoral immune response will be quantified by anti-glycoprotein E (anti-gE) antibody titers. Patients will receive two doses of RZV. Outcomes include seroconversion and geometric mean titers six weeks after completion of the vaccination schedule, persistence of antibody titers at one year, and incidence of confirmed herpes zoster during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosis of an autoimmune rheumatic disease (such as rheumatoid arthritis, systemic lupus erythematosus, axial spondyloarthritis, psoriatic arthritis, systemic sclerosis, Sjögren syndrome, idiopathic inflammatory myopathies, or primary systemic vasculitis) according to validated classification criteria.
* Clinical stability at the time of enrollment, defined as no change in disease-modifying therapy or corticosteroid dose in the preceding four weeks and no evidence of infection or disease flare.
* Current use of hydroxychloroquine or sulfasalazine in monotherapy for at least three months prior to inclusion.
* Can be under prednisone use of 5mg/week.
* Ability and willingness to comply with study procedures and follow-up visits.
* Provision of written informed consent.

Exclusion Criteria:

* Previous vaccination with recombinant zoster vaccine (RZV).
* History of herpes zoster or varicella infection within 12 months before enrollment.
* Concomitant use of systemic immunosuppressive therapy including but not limited to methotrexate, mycophenolate mofetil, azathioprine, cyclophosphamide, biologics, or JAK inhibitors.
* Use of glucocorticoids >5mg/week.
* Acute febrile illness or active infection at the time of vaccination.
* Pregnancy or breastfeeding.
* Known hypersensitivity to any component of the recombinant zoster vaccine.
* History of Guillain-Barré syndrome.
* Any condition that, in the investigators' judgment, could interfere with study participation or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of anti-glycoprotein E (anti-gE) antibodies six weeks after completion of the RZV vaccination schedule | Day 0 to six weeks after the second dose (Day 84)
  Humoral response will be assessed by ELISA quantification of anti-glycoprotein E antibodies. Seroconversion will be defined as a fourfold or greater increase from baseline or a fourfold increase above the lower limit of quantification for participants who are seronegative at baseline. The outcome is the proportion of participants who achieve seroconversion at Day 84.

SECONDARY OUTCOMES:
Geometric mean titers of anti-glycoprotein E antibodies six weeks after completion of the RZV vaccination schedule | Baseline (Day 0) and six weeks after the second dose (Day 84)
  Anti-glycoprotein E antibody concentrations will be measured in serum samples using an ELISA. Titers will be log-transformed and geometric mean titers will be calculated as the exponential of the mean of the log-transformed values. The outcome is the GMT at Day 84 and its change relative to baseline.
Persistence of antibody titers one year after completion of the RZV vaccination scheme | Day 0 to six weeks after the second dose (Day 84) and one year after the second dose (Day 365)
  Antibody persistence will be evaluated by quantifying anti-glycoprotein E antibody concentrations using ELISA. Results will be expressed as geometric mean titers obtained from log-transformed antibody levels. Seroconversion at one year will be defined as a fourfold or greater increase relative to baseline or a fourfold increase above the assay lower limit of quantification for participants seronegative at baseline.
Safety of RZV vaccine in ARD patients under immunomodulators | Day 0 to six weeks after the second dose (Day 84)
  Safety will be assessed by recording local and systemic adverse events through standardized diaries completed after each dose and confirmed during clinic visits. Events will be graded according to World Health Organization severity and CDC criteria.
Disease safety (flare) in ARD patients immunized with RZV | Day 0 to six weeks after the first dose (Day 42) and six weeks after the second dose (D84)
  Flare will be defined as a new flare or worsening of previous disease activity according to established scores for each ARD or the change of therapy. Disease activity will be evaluated in ARD patients according to specific standardized disease activity indexes: RA (DAS28 - Disease Activity Score 28, RA-CDAI - Rheumatoid Arthritis Clinical Disease Activity Index), SLE (SLEDAI2K - Systemic Lupus Erythematosus Disease Activity Index 2000), pSS (ESSDAI- EULAR Sjögren's Syndrome Disease Activity Index), IIM (MMT - Manual Muscle Test), AxS (ASDAS - Ankylosing Spondylitis Disease Activity Score), and vasculitis (Birmingham Vasculitis Activity Score).
Incidence of herpes zoster over one year following RZV vaccination in ARD patients under immunomodulators therapy | Day 42 (after the second dose) through one year after the second dose
  A suspected case of herpes zoster will be defined as (1) a new unilateral, dermatomal, rash with pain (broadly defined to include allodynia, pruritus, or other abnormal sensations) without any alternative diagnosis or (2A) or a vesicular rash suggestive of varicella zoster virus infection regardless of the distribution, and no alternative diagnosis; without any alternative diagnosis. For each suspected case, the rash will be photographed and samples will be collected from three lesions to confirm the diagnosis of HZ by real-time polymerase-chain reaction (PCR) assay. If the PCR results were indeterminate or if samples were not available, the final diagnosis will be determined by unanimous agreement among the five members of an ascertainment committee, which includes a dermatologist.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venerito V, Stefanizzi P, Cantarini L, Lavista M, Galeone MG, Di Lorenzo A, Iannone F, Tafuri S, Lopalco G. Immunogenicity and Safety of Adjuvanted Recombinant Zoster Vaccine in Rheumatoid Arthritis Patients on Anti-Cellular Biologic Agents or JAK Inhibitors: A Prospective Observational Study. Int J Mol Sci. 2023 Apr 9;24(8):6967. doi: 10.3390/ijms24086967. PMID 37108130
- [Background] Vink P, Delgado Mingorance I, Maximiano Alonso C, Rubio-Viqueira B, Jung KH, Rodriguez Moreno JF, Grande E, Marrupe Gonzalez D, Lowndes S, Puente J, Kristeleit H, Farrugia D, McNeil SA, Campora L, Di Paolo E, El Idrissi M, Godeaux O, Lopez-Fauqued M, Salaun B, Heineman TC, Oostvogels L; Zoster-028 Study Group. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine in patients with solid tumors, vaccinated before or during chemotherapy: A randomized trial. Cancer. 2019 Apr 15;125(8):1301-1312. doi: 10.1002/cncr.31909. Epub 2019 Feb 1. PMID 30707761
- [Background] Dagnew AF, Ilhan O, Lee WS, Woszczyk D, Kwak JY, Bowcock S, Sohn SK, Rodriguez Macias G, Chiou TJ, Quiel D, Aoun M, Navarro Matilla MB, de la Serna J, Milliken S, Murphy J, McNeil SA, Salaun B, Di Paolo E, Campora L, Lopez-Fauqued M, El Idrissi M, Schuind A, Heineman TC, Van den Steen P, Oostvogels L; Zoster-039 study group. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine in adults with haematological malignancies: a phase 3, randomised, clinical trial and post-hoc efficacy analysis. Lancet Infect Dis. 2019 Sep;19(9):988-1000. doi: 10.1016/S1473-3099(19)30163-X. Epub 2019 Aug 6. PMID 31399377
- [Background] Qian J, Lassere MN, Heywood AE, Liu B. Use of disease-modifying antirheumatic drugs and the subsequent risk of herpes zoster in older adults. Rheumatology (Oxford). 2021 Nov 3;60(11):5042-5051. doi: 10.1093/rheumatology/keab538. PMID 34508560
- [Background] Yun H, Yang S, Chen L, Xie F, Winthrop K, Baddley JW, Saag KG, Singh J, Curtis JR. Risk of Herpes Zoster in Autoimmune and Inflammatory Diseases: Implications for Vaccination. Arthritis Rheumatol. 2016 Sep;68(9):2328-37. doi: 10.1002/art.39670. PMID 26990731
- [Background] Yap RXL, Lai YW, Wei C, Ng JJW, Xu D, Feng S, Mu R, Thong BY, Xu C. Impact of Immunomodulatory Therapy on COVID-19 Vaccine Response in Patients with Autoimmune Inflammatory Rheumatic Diseases. Vaccines (Basel). 2024 Mar 6;12(3):274. doi: 10.3390/vaccines12030274. PMID 38543908
- [Background] van Sleen Y, van der Geest KSM, Huckriede ALW, van Baarle D, Brouwer E. Effect of DMARDs on the immunogenicity of vaccines. Nat Rev Rheumatol. 2023 Sep;19(9):560-575. doi: 10.1038/s41584-023-00992-8. Epub 2023 Jul 12. PMID 37438402